CLINICAL TRIAL: NCT00316641
Title: The Clinical Evaluation of Efficacy of Lipid-Lowing Tea on Hyperlipidemia Patients' Lipid Profiles
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: DMR93-IRB-71
Record Dates: First submitted 2006-04-20; First posted 2006-04-21 (Estimated); Last update posted 2006-11-07 (Estimated); Status verified 2006-03

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

INTERVENTIONS:
Drug: Lipid-lowing Tea

SUMMARY:
The purpose of this study is to determine whether the Lipid-lowing Tea is effective and safe in the treatment of Hyperlipidemia Patients

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 20-65 years;either sex
* Patient diagnosed with hyperlipidemia(fasting levels of TC>=200mg/dL),or TG>=200mg/dL but <400mg/dL,or LDL-C>=130mg/dL)
* Patient who has signed the informed consent form

Exclusion Criteria:

* Patient with pregnancy (or child bearing potential),or in lactation
* Patient with any lipid regulating agents within 4 weeks prior to study period
* Patient currently taking concomitant medications, such as oral contraceptives, or any medical treatment capable of interfering with lipid metabolism(eg thiazides, β-blockers, cyclosporins, itraconazole erythromycin,and danazol)
* Patient with medical history of hypothyroidism, pancreatitis, cholestasis, nephrotic syndrome, gall bladder disease, primary biliary cirrhosis.
* Patient with liver dysfunction (SGOT or SGPT>2x ULN)
* Patient with renal insufficiency (serum creatinine>1.3mg/dL)
* Patient with myocardial infarction,cerebrovascular disease,or major operations within 6 months prior to the study period.

Ages: 20 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Chia-I Tsai, V.S, Principal Investigator — China Medical University Hospital,Taichung,Taiwan
Locations (1):
- China Medical University Hospital, Taichung, Taiwan